CLINICAL TRIAL: NCT01934764
Title: Identification of Correlations Between Reaction to Biotine and Autoimmune Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, Assy Nimer, MD, Ziv Hospital
Other Study IDs: 0027-13-ziv
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-08

CONDITIONS: Autoimmune Disease
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- autoimmune disease

SUMMARY:
Working hypothesis and aims: Biotin is conjugated covalently to several proteins and use as a co-factor. Conjugation of biotin to non-targeted, unspecific proteins (e.g. immunoglobulins) leads to the breakage of the immune tolerance and to the formation of anti-biotin antibodies. Anti-biotin antibodies will be found in correlation with the progression and the present of autoimmune disease. In this research the correlation between immune response against biotin and the formations of autoimmune disease, will be studied:

A. Assessment of the possibility that biotin elicit immune response involved in the developmental stage of the autoimmune disease.

B. Assessment of the possibility that anti-biotin antibodies indicate the developmental stage of the autoimmune disease and therefore can serve as an disease early stage marker.

Methods: A. Patient recruitment. Gathering participant's medical record and blood samples. B. Records of clinical and biochemical measures. C. Serum of all patient will be tested for the correlation between biotin level, biotin bound to antibodies and anti-biotin antibodies to liver functions tests. D. Controlled test for repeatedly injected mice with biotinilated self-antibodies. Level of anti-biotin will be tested and their influence on the mouse. E. Determination of the correlation between biotinilated antibodies or anti-biotin antibodies to disease eruption or severance and autoimmune disease.

Expected results :Serum biotin-protein levels and Anti biotin antibodies levels are increased in patients with active autoimmune liver diseases.

Importance: The proof of connection between biotin-carrying immunoglobulins, anti biotin antibodies and autoimmune diseases will open new research direction of possible factors that cause to autoimmune disease.

Probable implications to Medicine: Identification of correlations between reaction to biotine and autoimmune diseases will enable their usage as biomarkers for autoimmune diseases, severity of the disease and personalization of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Freely given informed consent
* Autoimmune disease

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with autoimmune disease
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Biotin level Test | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical Center, Safed, Israel